CLINICAL TRIAL: NCT04336020
Title: The DETECT (Digital Engagement & Tracking for Early Control, & Treatment) Study
Brief Title: The DETECT(Digital Engagement & Tracking for Early Control, & Treatment) Study
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: CareEvolution Healthcare Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-20-7531
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Influenza; Virus
Keywords: Influenza; Viral infections; influenza-like illnesses (ILI); participant-reported outcomes (PRO); electronic health record (EHR)
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Develop an app-based nationwide study of individuals who routinely use a smartwatch or other wearable activity tracker to determine if individualized tracking of changes in heart rate, activity and sleep can provide an early indication of influenza-like illnesses (ILI) and possibly other viral infections.

DETAILED DESCRIPTION:
This study will be configured in CareEvolution's myDataHelps platform. This app-based platform will allow people to:

* Provide informed consent electronically
* Donate robust smartwatch and activity tracker data, as well as self-reported data.
* Sensor-collected data, which will vary between devices, but what is shared will always be entirely up to the participant. Investigators anticipate a minimum to include heart rate and activity, plus sleep duration when available.

  * This can include historical data collected by a sensor prior to the participants date of joining the study.
* Occasional survey-based participant-reported outcomes (PROs).
* Participant-entered physiologic data such as oral temperature
* Passively share environmental data such as air quality and weather that will be captured from external sources based on participants' "home" zip code. Optionally, if the participant consents to enable location/GPS services on their smartphone, higher grain environmental data will be enabled.
* Optionally connect to and share their electronic health record (EHR) data in the event they have an event that requires interaction with a health care provider

ELIGIBILITY:
Inclusion Criteria:

* Living in the U.S.
* 18 years or older
* Android or iPhone Smartphone user
* Any connected wearable (Apple Watch, Fitbit, Garmin watch connected to Apple Health or Google Fit, Amazfit)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators anticipate enrolling more than 100-thousand men and women in this study based on the inclusion criteria and otherwise no specific exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to study the individual heart rate, activity and sleep data in identifying influenza-like illnesses (ILI) in that individual using the CareEvolution's myDataHelps app-based platform. | Anticipated 2+-year duration of involvement in the study.
  The study will enable tens- to hundreds-of-thousands of interested smartwatch and active tracker wearers (e.g., Fitbit, Apple Watch, Garmin, Amazefit, OURA, Beddit, etc.) to donate their routinely collected data for research through a user-friendly app-based research platform to determine if individualized tracking of changes in heart rate, activity and sleep can provide an early indication of influenza-like illnesses (ILI) and possibly other viral infections.
  The study will capture timing, symptoms, and treatments of influenza-like illnesses (ILI) through on-app participant-reported outcome (PROs).
  When possible, use electronic health records (EHR) , available through in-app linkage, to supplement PRO-collected information about ILI or similar episodes.
  Data from optional devices (pulse ox, weight scales, BP cuffs, glucometers) may be integrated if the devices are connected and participant consents to share their data.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pandit, MD, Principal Investigator — Scripps Research Translational Institute
Locations (1):
- Scripps Research Translational Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The results of this research will be presented at meetings or in publication. However, the subject's identity will not be disclosed in those presentations.
Time Frame: Estimated 2025
Access Criteria: The results of this research will be presented at meetings or in publication.

REFERENCES:
- [Derived] Radin JM, Vogel JM, Delgado F, Coughlin E, Gadaleta M, Pandit JA, Steinhubl SR. Long-term changes in wearable sensor data in people with and without Long Covid. NPJ Digit Med. 2024 Sep 13;7(1):246. doi: 10.1038/s41746-024-01238-x. PMID 39271927
- [Derived] Quer G, Coughlin E, Villacian J, Delgado F, Harris K, Verrant J, Gadaleta M, Hung TY, Ter Meer J, Radin JM, Ramos E, Adams M, Kim L, Chien JW, Baca-Motes K, Pandit JA, Talantov D, Steinhubl SR. Feasibility of wearable sensor signals and self-reported symptoms to prompt at-home testing for acute respiratory viruses in the USA (DETECT-AHEAD): a decentralised, randomised controlled trial. Lancet Digit Health. 2024 Aug;6(8):e546-e554. doi: 10.1016/S2589-7500(24)00096-7. PMID 39059887